CLINICAL TRIAL: NCT05640037
Title: Urine Interleukin-37 as a Biomarker of Mortality Risk in Patients With Sepsis
Status: Completed | Type: Observational
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Dawei Wang
Record Dates: First submitted 2022-11-25; First posted 2022-12-07 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2023-12

CONDITIONS: Sepsis
Keywords: sepsis; interleukin-37; biomarker
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the efficacy of IL-37 as a biomarker to predict mortality risk in adults with sepsis.

DETAILED DESCRIPTION:
Sepsis patients admitted in the Department of Critical Care Medicine, Zhongnan Hospital will be included.

There are three groups of patients in this study: control group, sepsis group and septic shock group.

The interleukin-37 (IL-37) concentration in urine was analyzed in the day 1, 2, 4, 6.

Additionally, IL-37 concentration between blood stream infection groups and non-infection groups were analyzed. IL-37 concentration between survivors and non-survivors were also compared. IL-37 concentration were followed from day 1, 2, 4, 6.The correlation between the concentration of IL-37, IL-1β, IL-6、IL-10 and TNF-α were analyzed. Furthermore, the investigators will determine the correlation between the concentration of IL-37, sepsis associated organ dysfunction, 28-day mortality. Lastly, the predictive value of IL-37 to sepsis associated organ dysfunction and prognosis were explored.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Expected length of stay>24 hours in intensive care unit (ICU)
3. Sequential organ failure assessment (SOFA) score ≥ 2 on ICU admission with a suspicion of infection

Exclusion Criteria:

1. anuria
2. ICU readmission in 28 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ICU admission with a suspicion of infection
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
28-day all-cause mortality | 28 day
  Number of patients who were confirmed to be dead within 28-day from enrollment onto the study

SECONDARY OUTCOMES:
ICU all-cause mortality | 28 day
  Number of patients who were confirmed to be dead in ICU from enrollment onto the study
ICU length of stay | 28 day
  Length of intensive care unit stay
Hospital length of stay | 28day
  Length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Dawei Wang, MD, Study Chair — Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No